CLINICAL TRIAL: NCT01835379
Title: A Randomized, Open Label Controlled Trial of OASIS® Ultra Tri-Layer Matrix Compared to Standard Care in the Healing of Diabetic Foot Ulcers
Brief Title: Study of Oasis Ultra in Diabetic Foot Ulcers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Healthpoint (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 815-999-09-010
Record Dates: First submitted 2013-04-16; First posted 2013-04-18 (Estimated); Results first posted 2015-01-22 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetes; Diabetic Foot Ulcer; Diabetic Foot Wound; Non-healing foot wound; Oasis; Diabetic neuropathy
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Diabetic Neuropathies | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oasis (Experimental): Oasis
  Interventions: Device: Oasis
- Standard (Other): Standard Care
  Interventions: Other: Standard

INTERVENTIONS:
Device: Oasis — Oasis Ultra will be applied once per week for up to 12 weeks.
  Arms: Oasis
Other: Standard
  Other Names: Standard Care
  Arms: Standard

SUMMARY:
Many people with diabetes will develop a non-healing diabetic foot ulcer. Many ways are available to try to get a diabetic foot ulcer to heal, including application of Oasis Ultra. The hypothesis to be tested is that application of Oasis Ultra will cause more diabetic foot ulcers to heal than wounds treated with regular medical care. Subjects will have their diabetic foot wounds treated for up to 12 weeks with Oasis Ultra or regular medical care .

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent, which will consist of reading, signing, and dating the informed consent document after the Investigator, sub-Investigator or other designated study staff member has explained the study procedures, risks, and contact information.
* Subjects 18 years of age or older of either sex with a history of diabetes mellitus (Type 1 or 2) requiring medication (insulin and/or oral/injectable) to control blood glucose levels.
* A non-healing, Wagner grade 1 or 2, neuropathic diabetic foot ulcer.
* Willing and able to make all required study visits.
* Able to follow instructions.
* An ulcer present on any part of the plantar surface of the foot, which is 0.5 cm2 to 10 cm2 (inclusive), as measured at the Screening Visit prior to debridement, with a duration ≥ 6 weeks (documented in the patient's history or by patient report of onset) but not more than 12 months.
* Separation of at least 5 cm (wound edge to wound edge) if ≥ 2 wounds are present.
* Adequate arterial blood flow as evidenced by an ankle brachial index (ABI) of > 0.7 and ≤ 1.1. If the ABI is greater than 1.1, then a toe pressure of > 40 mmHg OR a transcutaneous oxygen pressure (TcPO2) ≥ 40 mmHg must be present. Either toe pressure or TcPO2 is also acceptable in lieu of ABI, but if both are obtained, each must meet its respective cutoff.

Alternatively, a Doppler waveform consistent with adequate flow to the region of the foot with the target ulcer (biphasic or triphasic waveforms) is acceptable (test result must be included in the source document).

* Target ulcer is not infected based on clinical assessment.
* Able to perform any required dressing changes at home or have a caregiver who can perform the dressing changes.
* Willing to use an appropriate off-loading device to keep weight off of foot ulcers.
* Blood counts and blood chemistry values as follows:

  * Alanine aminotransferase (ALT) ≤ 3x upper limit of normal
  * Aspartate aminotransferase (AST) ≤ 3x upper limit of normal
  * Serum albumin ≥ 2.0 g/dL •Pre-albumin levels of ≥ 10 mg/dL
  * Alkaline phosphatase ≤ 500 U/L •Serum total bilirubin ≤ 3.0 mg/dL
  * Serum BUN < 75 mg/dL •Serum creatinine ≤ 4.5 mg/dL
  * HbA1c ≤ 12% •Hemoglobin (Hgb) > 8.0 g/dL
  * WBC > 2.0 x 109/L •Absolute neutrophil count > 1.0 x 109/L
  * Platelet count > 50 x 109/L

Exclusion Criteria:

* Contraindications or hypersensitivity to the use of the study device or its components (e.g., porcine sensitivity).
* Participation in another investigational study within thirty (30) days of Visit 1 or planned participation overlapping with this study.
* Subjects with evidence of gangrene on either lower limb.
* Ulcers that require negative pressure or hyperbaric oxygen therapy.
* The Medical Monitor may declare any subject ineligible for a valid medical reason.
* Current treatment with disallowed medications or therapies. Subjects may not be enrolled into the study while using systemic antibiotics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2013-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert B Slade, MD, Study Chair — Healthpoint
Locations (15):
- United States (15):
  - Little Rock, Arkansas
  - Carlsbad, California
  - Fair Oaks, California
  - Fresno, California
  - San Diego, California
  - Evansville, Indiana
  - Madisonville, Kentucky
  - Shreveport, Louisiana
  - Saginaw, Michigan
  - Bayonne, New Jersey
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - McAllen, Texas
  - Virginia Beach, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Oasis: Oasis
  Oasis Ultra applied once per week for up to 12 weeks.
- Standard: Standard Care
  Standard Care as chosen by the Investigator
Period: Overall Study
Arm/Group | Oasis | Standard
Started | 41 | 41
Completed | 41 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oasis | Standard | Total
Number analyzed (Participants) | 41 | 41 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (10.9) | 56.6 (10.8) | 56.9 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 32 | 30 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 16 | 26
  Not Hispanic or Latino | 31 | 25 | 56
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 6 | 12
  White | 33 | 33 | 66
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 41 | 41 | 82
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 32.9 (8.9) | 33.6 (6.1) | 33.3 (7.6)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Wounds Closed
Time Frame: At the end of 12 Weeks
Measure: Number; unit: percentage of wounds closed
Arm/Group | Oasis | Standard
Number analyzed (Participants) | 41 | 41
percentage of wounds closed | 54 | 32

2. Secondary Outcome: Time to Wound Closure
Description: Kaplan-Meier (K-M) analysis was employed to estimate the median time in weeks to complete ulcer closure.
Time Frame: During the 12 Week treatment period
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Oasis | Standard
Number analyzed (Participants) | 41 | 41
weeks | 9 [1.0 to 12.0] | 11 [1.0 to 12.0]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the 12-week treatment period.
Arm/Group | Oasis | Standard
Serious Adverse Events (participants affected / at risk) | 10/41 | 10/41
Other Adverse Events (participants affected / at risk) | 0/41 | 0/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oasis (N=41) | Standard (N=41)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 2 (2) | 0 (0)
Osteomyelitis (Infections and infestations) | 2 (2) | 5 (5)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lower GI hermorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
GERD (Gastrointestinal disorders) | 0 (0) | 1 (1)
Transient ischemic attack (TIA) (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release.